CLINICAL TRIAL: NCT00034710
Title: A Double-Blind Controlled Pilot Study of High-Dose Capsaicin Patches in the Treatment of Pain Associated With Postherpetic Neuralgia
Brief Title: Pilot Study of High-Dose Capsaicin Patches to Treat Postherpetic Neuralgia Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeurogesX (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: C102
Record Dates: First submitted 2002-05-01; First posted 2002-05-02 (Estimated); Last update posted 2006-02-07 (Estimated); Status verified 2006-02

CONDITIONS: Neuralgia; Pain; Peripheral Nervous System Diseases; Herpes Zoster
Keywords: Analgesics/*therapeutic use; Capsaicin/*administration & dosage/adverse effects; Herpes Zoster/*complications/drug therapy; Neuralgia/*drug therapy/etiology; Pain; Capsicum; Pepper; Dermal assessment; Pain measurement; Diary; PHN; Postherpetic Neuralgia; allodynia; hyperalgesia; shingles; varicella
MeSH Terms: conditions — Neuralgia; Pain; Peripheral Nervous System Diseases; Herpes Zoster; Neuralgia, Postherpetic; Hyperalgesia; Chickenpox

INTERVENTIONS:
Drug: Capsaicin Patch

SUMMARY:
The purpose of this study is to gain initial information on the tolerability of high-dose capsaicin patches in patients with Painful Postherpetic Neuralgia. The study will also collect preliminary information on safety and efficacy.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

Patients may be eligible for this study if they:

* Have a diagnosis of Painful Postherpetic Neuralgia and are at least 6 months post vesicle crusting.
* Are in good health.
* Have an adequate pain score during the screening period.
* Have painful areas (maximum of two sites) below the neck.
* If female, are of non-childbearing ability as defined by absence of menses for a minimum of 3 months or surgically sterile.
* If male, are willing to agree to take adequate birth control precautions with their partner for 60 days following experimental drug exposure.
* Have unbroken skin with good perfusion over the painful area(s).
* Have the ability to feel capsaicin-mediated sensations, as evidenced by ability to feel topically applied OTC capsaicin cream.
* Are on a stable and continuous medication regimen, with no change in dosage for 21 days prior to study start, and are willing to maintain concomitant medications at current doses throughout the study.
* Are willing and able to use oral opioid-based analgesic agents for relief, in case this is needed to relieve acute pain associated with the application of capsaicin patches.
* Are 18 years of age or older.
* Are willing and able to comply with the protocol

Exclusion Criteria:

Patients will not be eligible for this study if they:

* Have diffusely distributed neuropathic pain (i.e., pain that is evident in more than 2 different sites). Subjects must not have significant pain outside the areas to be treated.
* Have any implanted medical device (spinal cord stimulator, intrathecal pump or peripheral nerve stimulator) for the treatment of neuropathic pain.
* Currently (within the past 21 days) use topically applied non-steroidal anti-inflammatory drugs, local anesthetics, steroids or capsaicin products on the painful areas.
* Currently (within the past 21 days) use topical agents such as lidoderm patch 5%, topical steroids or aspirin.
* Have a history or current problem with prescription drug or illicit substance abuse (from self report or as judged by investigator).
* Currently have an abuse problem with alcohol (from self-report or as judged by investigator).
* Are suspected of psychosocial gain/benefit of continued pain as judged by the investigator or primary treating physician.
* Plan to travel more than 100 miles from home during the study or engage in unusual activities that might exacerbate pain.
* Have poor cardiac, renal, hepatic, or pulmonary function judged by the investigator or primary treating physician.
* Have a laboratory value at screening outside the normal range, unless it is judged by the investigator as not clinically significant after appropriate evaluation.
* Have hypersensitivity to capsaicin (i.e., chili peppers or OTC capsaicin products), local anesthetics, oral opioid-based analgesic agents, or adhesives.
* Have a high tolerance to opioids.
* Currently using Class 1 anti-arrhythmic drugs (such as tocainide and mexiletine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2002-03; Study Completion 2002-10

CONTACTS AND LOCATIONS:
Overall Officials: John A Jermano, Study Director — NeurogesX
Locations (8):
- United States (8):
  - Arizona Research Center, Phoenix, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Anchor Research Center, Naples, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Brigham and Women's Hospital, Pain Trials Center, Boston, Massachusetts
  - University of Utah Pain Management Center, Salt Lake City, Utah
  - University of Wisconsin Hospital, Neurology Department, Madison, Wisconsin